CLINICAL TRIAL: NCT05222932
Title: A Phase I Open-Label, Dose-escalation Clinical Trial of Tumor Necrosis Factor Alpha and IL-2 Coding Oncolytic Adenovirus TILT-123 and Avelumab in Solid Tumor Patients (Melanoma and SCCHN) Refractory to or Progressing After Anti-PD(L)1
Brief Title: Oncolytic Adenovirus TILT-123 and Avelumab for Treatment of Solid Tumors Refractory to or Progressing After Anti-PD(L)1
Acronym: AVENTIL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TILT Biotherapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILT-T776
Record Dates: First submitted 2022-02-01; First posted 2022-02-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Head and Neck Squamous Cell Carcinoma
Keywords: oncolytic virus; immunotherapy; immune checkpoint inhibitor
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck | interventions — Tumor Necrosis Factor-alpha; avelumab

STUDY DESIGN:
Intervention Model Description: open-label, single arm, dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TILT-123 and avelumab (Experimental): Patients will receive multiple administrations of TILT-123 and avelumab.
  Escalation to the next dose of TILT-123 level will occur when the safety data has been evaluated for all patients in the preceding dose level.
  Interventions: Biological: TILT-123; Drug: Avelumab

INTERVENTIONS:
Biological: TILT-123 — TNFalpha and IL-2 coding oncolytic adenovirus TILT-123
  Other Names: TNFalpha and IL-2 coding oncolytic adenovirus TILT-123; Ad5/3-E2F-d24-hTNFa-IRES-hIL2
Drug: Avelumab — Anti-PDL1 antibody
  Other Names: anti-PD-L1 monoclonal antibody

SUMMARY:
This is a phase 1, dose-escalation trial evaluating the safety of oncolytic adenovirus TILT-123 in combination with avelumab in patients with advanced solid tumors refractory to or progressing after anti-PD(L)1.

DETAILED DESCRIPTION:
This is an open-label, phase 1, dose-escalation trial evaluating the safety of TILT-123 TILT-123 in combination with avelumab in patients with advanced solid tumors (SCCHN and melanoma) refractory to or progressing after anti-PD(L)1. TILT-123 is an oncolytic adenovirus coding for tumor necrosis factor alpha and interleukin 2. The trial is conducted in Helsinki (Finland).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be over 18 years of age
2. Subject must have pathologically confirmed refractory or recurrent injectable solid tumor (melanoma or SCCHN), which cannot be treated with curative intent with available therapies and is refractory to or progressing after anti-PD(L)1 immunotherapy.
3. Standard therapy has failed, it does not exist, is not available or is unlikely to result in meaningful clinical benefit (as assessed by the investigator). Multiple prior therapies (eg. surgery, chemotherapy, radiation, checkpoint inhibitors, kinase inhibitors, biological therapies) are allowed.
4. At least one tumor lesion of 15 mm or bigger must be available for biopsy and injections that, in the opinion of the investigator, is accessible to repeated injections and biopsies without major safety concerns.
5. The disease burden must be evaluable, but does not need to fulfil RECIST 1.1
6. Patients must have received at least 6 weeks of prior PD-1/PDL-1 blocking antibody therapy (e.g. 3x 2w cycle or 3x 3w cycle) within the past up to 12 months
7. Patients must have experienced unequivocally documented radiographic progression of disease during or within 6 weeks after the last dose of such treatment.
8. Subject must have adequate hepatic and renal functions, including the following laboratory parameters:

   1. Platelets > 75 000/mm3
   2. Haemoglobin ≥ 100 g/L.
   3. AST and ALT < 3 x ULN.
   4. GFR >60 ml/min (Cockcroft-Gault formula).
   5. Leukocytes (WBC) > 3,0
   6. Bilirubin <1,5 x ULN
9. Men and women must be willing to use adequate forms of contraception from screening, during the trial, and for a minimum of 90 days after end of treatment, in accordance with the following:

   1. Women of childbearing potential: Barrier contraceptive method (i.e. condom) must be used in addition to one of the following methods: Intrauterine device or hormonal contraception (oral contraceptive pills, implant, transdermal patches, vaginal ring or long-acting injections).
   2. Women not of childbearing potential: Barrier contraceptive method (i.e. condom) must be used.
   3. Men: Barrier contraceptive method (i.e. condom) must be used.
10. Subject must demonstrate a WHO/ECOG performance score of 0-1
11. Subject must have life expectancy longer than 3 months according to investigator assessment
12. Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent approved by the Independent Ethics committee prior to the initiation of any screening or study -specific procedure.

Exclusion Criteria:

1. Prior organ transplantation including allogenic stem-cell transplantation or subject is using systemic immunosuppressive medications (eg. corticosteroids or drugs used in treatment of autoimmune disease). Exempted are the following which can be allowed at screening and during the trial: a) replacement corticosteroids if e.g. the patient has adrenal insufficiency after prior immunotherapy b) inhaled and topical treatments c) up to 20 mg/d of prednisone/prednisolone (or equivalent).
2. Treated with any anti-cancer therapy within 30 days prior to the first virus injection. Anti-cancer therapy is defined as anti-cancer agents (e.g. cytotoxic chemotherapy, immunotherapy, signal-transduction inhibitors, biological therapies) and investigational agents. An investigational agent is any drug or therapy that is currently not approved for use in humans. Continuation of bone modifying agents (eg. bisphosphonate or denosumab) is allowed if started at least 3 months before. Palliative radiation is not allowed within 14 days of the first virus injection (before or after), but it is allowed after day 15 during the trial treatment period, if deemed necessary by the investigator.
3. Subject has a history of another active invasive cancer within the past 5 years, except curatively treated basalioma or squamous cell carcinoma of the skin
4. Clinically significant (i.e. active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
5. Subject has a history of interstitial parenchymal lung disease.
6. Subject has a LDH value > 3 x ULN (melanoma)
7. Subject has a history of severe hepatic dysfunction, hepatitis, HIV or other severe chronic but active infectious diseases requiring systemic therapy, e.g. tuberculosis
8. Subject is using proton pump inhibitors or antibiotics during screening period
9. Subject has a history of a coagulation disorder or abnormality in coagulation parameters, as defined by an international normalized ratio not within the normal range, or has received oral or parenteral anticoagulants or thrombolytic agents for therapeutic or prophylactic purposes (including coumadin and warfarin) within 10 days of the first dose of the study treatments. Low molecular weight heparin is permitted if the international normalized ratio is within the normal range
10. Any other medical condition or laboratory abnormality that in the judgment of the principal investigator, may increase the risk associated with study participation or may interfere with interpretation of study results and /or otherwise make the patient inappropriate for entry into this trial.
11. Subject is pregnant, breastfeeding or intend to become pregnant
12. Subject has untreated brain metastases. Treated and asymptomatic brain metastases which have not progressed in 3 months prior to study entry are allowed.
13. Any known or suspected allergy to TILT-123 or ingredients present in the drug product as listed in this protocol.
14. Any known or suspected allergy to avelumab or ingredients present in the drug product as listed in summary of product characteristics (SmPC), including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE Grade ≥ 3).
15. Known current alcohol or drug abuse
16. Vaccination with live vaccines in the past 30 days prior to start of investigational treatment
17. History of immune-related adverse events to previous immunotherapy which led to discontinuation from treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with any (serious and non-serious) Adverse Events. | 85 days
  Safety I
Number of Participants with abnormal laboratory values. | 85 days
  Safety II
Number of Participants with vital sign abnormalities. | 85 days
  Safety III
Number of Participants with Adverse Events assessed by 12- lead electrocardiograms (ECGs) | 85 days
  Safety IV

CONTACTS AND LOCATIONS:
Overall Officials: Tuomo Alanko, Principal Investigator — Docrates Cancer Center
Locations (2):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Docrates Cancer Center, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No